CLINICAL TRIAL: NCT06844851
Title: Evaluation of Genetic-molecular Causes of Out-of-Hospital Cardiac Arrest: from Patients to Families
Acronym: GenetiCA
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Enrico Baldi, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: GenetiCA
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Cardiac Arrest (CA)
Keywords: Out-of-hospital cardiac arrest; genetic; cardiovascular diseases
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- OHCA patients under 50 years: All the patients suffering from OHCA of medical etiology in Lombardy Region ≤50 years, for whom resuscitation manoeuvres was started by EMS (AREU)

SUMMARY:
The aims are to define the exact prevalence of hereditary heart diseases in out-of-hospital cardiac arrest (OHCA) patients taking also into account gender, patient and OHCA characteristics, provincial settings and environmental pollution; to stratify the individualized arrhythmic risk of proband's family members to prevent further sudden cardiac deaths; to refine the classification of the variants of uncertain significance (VUS) on genes which can have the capability to drive to molecular alterations leading to arrhythmogenic hereditary heart diseases. A blood sample will be obtained during resuscitation from all the patients aged ≤50 years suffering an OHCA in Lombardy Region and then analysed for genetic variants possibly causative of cardiac diseases. Genetic data will be merged with patient, OHCA and post-resuscitation data thanks to the connection with LombardiaCARe, whilst pollution data will be retrieved from ARPA Lombardia for free. A genetic counselling and clinical-instrumental evaluation of the proband's first-degree family members will be performed if a pathogenic/likely pathogenic variant or a VUS will be disclosed during the genetic analysis.

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest (OHCA) is one of the most important causes of death and the majority of OHCAs are attributable to cardiovascular diseases. The proportion of young patients (aged ≤ 50 years) among the OHCA victims is not negligible (1-20 per 100.000 inhabitants). Many OHCAs in this population could be due to alterations to genes leading to molecular alterations causing arrhythmogenic diseases. That's why, other than performing an autopsy in all unexplained deaths in young people (≤50 years), it is recommended by the major European and American scientific societies to perform a post-mortem genetic test for the most common genes associated with rare arrhythmogenic hereditary heart diseases through 5-10 mL of whole blood preserved in EDTA. Such procedures, however, are not routinely performed and usually they are performed only on hospitalized patients who, unfortunately, represents a minority of OHCA victims. The execution of a post-mortem genetic test can in fact explain up to 15-25% of sudden cardiac deaths in young people and for this reason a joint consensus document among 5 scientific societies stresses that sudden death in young people should be considered a public health priority given the high percentage of inherited genetic heart diseases and the impact on the family, encouraging the investment of public funds in research in this field. A number of studies evaluating arrhythmogenic cardiac disease in patients who survived or died from cardiac arrest have been performed over the past 2 decades. In some of them, carried out in the early 2000s, researchers focused their analysis on genes related to long QT syndrome (LQTS) and catecholaminergic polymorphic ventricular tachycardia (CPVT), finding pathogenic variants in 11-40% of patients. In more recent years, thanks to the use of new techniques such as next-generation sequencing (NGS), it has been possible to extend the analysis, with optimisation of costs and genetic material required, to multi-gene panels exploring genes linked to LQTS, CPVT, short QT syndrome (SQTS), Brugada syndrome (BrS), arrhythmogenic cardiomyopathy (ACM), hypertrophic cardiomyopathy (HCM), restrictive cardiomyopathy (RCM), dilated cardiomyopathy (DCM) and non-compaction cardiomyopathy (LCVN). However, all these studies to date involved a limited number of patients, selected either from survivors of OHCA or from victims of OHCAs for whom autopsy findings were required. Moreover, these studies focused on limited geographic areas. There are currently no studies that homogeneously and cross-sectionally involve an entire geographic area by evaluating all patients who suffer from an OHCA in that territory.

All the patients suffering from OHCA of medical etiology in Lombardy Region ≤50 years, for whom resuscitation manoeuvres was started by EMS (AREU), will be enrolled. The EMS personnel will store 10 mL of blood acquired during resuscitation manoeuvres through the vascular access routes positioned for patient's care. This will not alter the standard patient treatment. The blood will be stored at 4°C in the EMS provincial stations and will be periodically collected. The EMS personnel will acquire informed consent for genetic analysis by a third party belonging to the same genetic line as the patient or will ask for a contact address for subsequent contact by the research team.

The laboratory will perform aliquoting and genetic analysis. The DNA extraction will be performed through an automated extractor and the extracted DNA samples will be sequenced using 1. An updated customized Agilent panel including known and validated disease genes as well as novel candidate genes; 2. the Illumina TrusightCardio multi-gene panel, including all genes most commonly associated with LQTS, CPVT, SQTS, BrS, ACM, HCM, RCM, DCM, RASopathies, lysosomal storage diseases, other rare genetic cardiovascular diseases, rare forms of autosomal recessive myopathies and heritable metabolic diseases.

In case of a P-LP variant or a VUS was identified, genetic counselling and clinical-instrumental evaluation of the proband's first-degree family members will be offered at the Fondazione IRCCS Policlinico San Matteo. All the family members will be screened with an electrocardiogram and an echocardiogram, and the need for execution of other diagnostic tests will be evaluated based on individual characteristics and the family history of each patient. Moreover, if a P-LP variant was identified in the proband, the first-degree family members will be invited to undergo a genetic test to verify if they are carriers of the same variant. All the data regarding the therapeutic actions performed to prevent further sudden cardiac deaths will be collected.

For each patient data regarding the pre-hospital OHCA characteristics, the treatment, the post-resuscitation clinical and laboratory data (for survived patients) and the survival will be collected using the LombardiaCARe. Data regarding the genetic analysis and, concerning the family members, all the data regarding the past medical history and the diagnostic and therapeutic procedures performed will be collected. All these data will be filed using the REDCap® (Research Electronic Data Capture) platform, hosted at Fondazione IRCCS Policlinico San Matteo, and will be merged into a unique database.

The variant prevalence will be calculated as the ratio of patients in whom a variant is found to the total number of patients with OHCA and its binomial exact 95% confidence interval. Moreover, the differences in the prevalence of P/LP or VUS in patients stratified for gender, province, presenting rhythm and other OHCA characteristics will be compared. The difference in survival at hospital arrival and at discharge between patients with or without a potential P-LP variant will be computed. Finally, differences in prevalence and survival according to the level of pollutants in the different geographical areas will be properly evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All the patients suffering from OHCA of medical etiology in Lombardy Region ≤50 years, for whom resuscitation manoeuvres was started by EMS (AREU)

Exclusion Criteria:

* Patients under 18 years old
* Patients with a non-medical cause of the cardiac arrest

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All the patients suffering from OHCA of medical etiology in Lombardy Region ≤50 years, for whom resuscitation manoeuvres was started by EMS (AREU)
Sampling Method: Non-Probability Sample
Enrollment: 1725 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of pathogenic/likely-pathogenic variants | December 2027
  Percentage of patients with pathogenic/likely-pathogenic variants or with variants of unknown significance (VUS) as defined by ACMG guidelines out of the total number of patients analysed

SECONDARY OUTCOMES:
Familiar screening | December 2027
  Number of families and family members who received clinical-instrumental evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No